CLINICAL TRIAL: NCT02663453
Title: Effectiveness of Multicomponent Lipid Emulsion in Preterm Infants Requiring Parenteral Nutrition: A Two-Center, Double-Blind Randomized Clinical Trial
Brief Title: Effectiveness of Multicomponent Lipid Emulsion in Preterm Infants Requiring Parenteral Nutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Dr Wilaiporn Techasatid, Head of Neonatology, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-PE-1-033/56
Record Dates: First submitted 2016-01-11; First posted 2016-01-26 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Cholestasis
Keywords: preterm; parenteral nutrition; cholestasis; fish oil
MeSH Terms: conditions — Cholestasis; Premature Birth; Hyperphagia | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): multicomponent lipid emulsion composed of 30% soybean oil, 30% MCTs, 25% olive oil and 15% fish oil (SMOF lipid) was administered at a dose of 1gm/kg/day within 24 hours after birth; lipid dosage was increased by an increment of 0.5 gm/kg/day until the maximal dose of 3.5 gm/kg/day was reached.The macronutrients and micronutrients were provided using the same products in both groups.
  Interventions: Drug: multicomponent lipid emulsion
- control group (Active Comparator): pure soybean oil lipid emulsion(intralipid) was administered at a dose of 1gm/kg/day within 24 hours after birth; lipid dosage was increased by an increment of 0.5gm/kg/day until the maximal dose of 3.5gm/kg/day was reached.The macronutrients and micronutrients were provided using the same products in both groups.
  Interventions: Drug: pure soybean oil lipid emulsion

INTERVENTIONS:
Drug: multicomponent lipid emulsion — Lipids were first administered at a dose of 1gm/kg/day within 24 hours after birth for both groups; lipid dosage was increased by an increment of 0.5 gm/kg/day until the maximal dose of 3.5 gm/kg/day was reached.
  Other Names: SMOF lipid
  Arms: study group
Drug: pure soybean oil lipid emulsion — Lipids were first administered at a dose of 1gm/kg/day within 24 hours after birth for both groups; lipid dosage was increased by an increment of 0.5 gm/kg/day until the maximal dose of 3.5 gm/kg/day was reached.
  Other Names: Intralipid
  Arms: control group

SUMMARY:
The purpose of this study is to compare the effects of a multicomponent lipid emulsion containing 30% soybean oil, 30% medium-chain triglycerides, 25% olive oil, and 15% fish oil with a conventional pure soybean oil lipid emulsion on the incidence of neonatal cholestasis, infant growth, infant morbidity and the biochemical assessment of liver enzymes.

DETAILED DESCRIPTION:
Intravenous lipid emulsions are the major sources of non-protein energy and provision of required essential fatty acids.

The reference lipid emulsion, widely used for many years, is prepared from soybean oil, which is rich in omega 6 polyunsaturated fatty acids and phytosterols that contribute to hepatotoxicity and their metabolites result in pro-inflammatory eicosanoid production.

Existing evidence strongly supports a pathogenetic role of inflammation and oxidative stress on parenteral nutrition associated liver disease.

Subsequent development of lipid emulsions has focused on reducing the amount of soybean oil and replacing it with other oils.Moreover the omega 3 fatty acids from fish oil are metabolized to anti-inflammatory eicosanoids which can prevent inflammatory responses.

A novel multicomponent lipid emulsion may prevent liver injury, improve growth and decrease morbidity in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants with a gestational age of less than 30 weeks
* Who required parenteral nutrition for at least 7 days

Exclusion Criteria:

* Evidence of congenital infection
* Perinatal asphyxia
* Congenital anomalies
* Severe IVH
* Thrombocytopenia
* Shock or circulation failure
* Renal or hepatic disorders.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilaiporn Techasatid, doctor, Principal Investigator — Department of Pediatrics, Faculty of Medicine, Thammasat University, 95 Paholyothin Road, Klongluang, Pathumthani, 12120 Thailand.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tomsits E, Pataki M, Tolgyesi A, Fekete G, Rischak K, Szollar L. Safety and efficacy of a lipid emulsion containing a mixture of soybean oil, medium-chain triglycerides, olive oil, and fish oil: a randomised, double-blind clinical trial in premature infants requiring parenteral nutrition. J Pediatr Gastroenterol Nutr. 2010 Oct;51(4):514-21. doi: 10.1097/MPG.0b013e3181de210c. PMID 20531018
- [Result] Rayyan M, Devlieger H, Jochum F, Allegaert K. Short-term use of parenteral nutrition with a lipid emulsion containing a mixture of soybean oil, olive oil, medium-chain triglycerides, and fish oil: a randomized double-blind study in preterm infants. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1 Suppl):81S-94S. doi: 10.1177/0148607111424411. PMID 22237883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled preterm infants who required parenteral nutrition for at least 7 days from 2 academic medical centers in Bangkok. The last patient completed in December 2015
Groups:
- Study Group: multi component lipid emulsion composed of 30% soybean oil, 30% MCTs, 25% olive oil and 15% fish oil (SMOF lipid) was administered at a dose of 1 gm/kg/day within 24 hours after birth; lipid dosage was increased by an increment of 0.5 gm/kg/day until the maximal dose of 3.5 gm/kg/day was reached.The macro nutrients and micro nutrients were provided using the same products in both groups. Parenteral lipid was temporarily stopped when plasma triglyceride (TG) concentrations exceeded 250 mg/dL. Minimal enteral feeding was initiated on the day of birth and intake was advanced with 20 ml/ kg/day of breast milk or preterm formula. Parenteral nutrition was stopped when the oral feeding reached 120 ml/kg/day
- Control Group: pure soybean oil lipid emulsion was administered at a dose of 1 gm/kg/day within 24 hours after birth; lipid dosage was increased by an increment of 0.5 gm/kg/day until the maximal dose of 3.5gm/kg/day was reached.The macronutrients and micronutrients were provided using the same products in both groups.
  Parenteral lipid was temporarily stopped when plasma triglyceride (TG) concentrations exceeded 250 mg/dL. Minimal enteral feeding was initiated on the day of birth and intake was advanced with 20 ml/ kg/day of breast milk or preterm formula. Parenteral nutrition was stopped when the oral feeding reached 120 ml/kg/day
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 22 | 22
Completed | 17 | 18
Not Completed | 5 | 4
Not completed — Death | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 27.6 (2.2) | 28.4 (1.2) | 28.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Thailand | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Neonatal Cholestasis
Description: direct bilirubin level of more than 2 mg/dL
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
Participants | 1 | 2

2. Secondary Outcome: Neonatal Morbidities
Description: retinopathy of prematurity, bronchopulmonary dysplasia
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
Participants
  retinopathy of prematurity | 7 | 6
  bronchopulmonary dysplasia | 10 | 9

3. Secondary Outcome: Incidence of Extrauterine Growth Restriction (EUGR)
Description: weight that is less than the tenth percentile for corrected gestational age by the time of discharge
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
Participants | 8 | 12

4. Secondary Outcome: Weight Gain
Description: in-hospital weight gain at birth until discharge (gram/day)
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: gram/day
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
gram/day | 19.7 (3.9) | 18.8 (3.9)

5. Secondary Outcome: Height Gain
Description: in-hospital height gain at birth until discharge (cm/week)
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
cm/week | 0.9 (0.2) | 0.8 (0.2)

6. Secondary Outcome: Head Circumference Gain
Description: in-hospital head circumference gain at birth until discharge (cm/week)
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
cm/week | 0.7 (0.2) | 0.7 (0.2)

7. Secondary Outcome: Assessment of Gamma Glutamyltranspeptidase (GGT)
Description: blood samples were obtained before enrollment, week 1, 2 and 3 (U/L) after parenteral nutrition administration
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
U/L
  before enrollment | 134.7 (113.8) | 138.7 (62.6)
  week 1 | 73.8 (58.8) | 79.5 (45.4)
  week 2 | 63.1 (47.5) | 68.6 (43.5)
  week 3 | 94.0 (68.3) | 95.4 (85.2)

8. Secondary Outcome: Assessment of Alanine Aminotransferase (ALT)
Description: blood samples were obtained before enrollment, week 1, 2 and 3 (U/L) after parenteral nutrition administration
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
U/L
  before enrollment | 16.3 (12.8) | 15.1 (7.1)
  week 1 | 14.7 (7.8) | 15.1 (7.2)
  week 2 | 17.1 (8.7) | 19.8 (13.3)
  week 3 | 17.5 (6.8) | 17.7 (7.9)

9. Secondary Outcome: Assessment of Aspartate Aminotransferase (AST)
Description: blood samples were obtained before enrollment, week 1, 2 and 3 (U/L) after parenteral nutrition administration
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 22 | 22
U/L
  before enrollment | 61.8 (21.6) | 55.6 (28.1)
  week 1 | 26.5 (22.0) | 26.0 (9.6)
  week 2 | 26.2 (8.0) | 24.4 (6.2)
  week 3 | 24.2 (3.7) | 25.9 (8.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/22 | 4/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No